CLINICAL TRIAL: NCT04760353
Title: The Effect of a Probiotic Mixture on the Symptoms and Fecal Microbiota in Obese Patients With Irritable Bowel Syndrome, Randomised, Double-blind, Controlled Study
Brief Title: The Effect of a Probiotic Mixture in Obese Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Rijeka (Other)
Collaborators: Institute AllergoSan (Unknown)
Responsible Party: Principal Investigator, Goran Hauser, Clinical Professor, University Hospital Rijeka
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Omni Stress 1.1
Record Dates: First submitted 2021-01-26; First posted 2021-02-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: IBS - Irritable Bowel Syndrome; Obesity
Keywords: IBS; Obesity; microbiota
MeSH Terms: conditions — Irritable Bowel Syndrome; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): one powder portion bag of the probiotic mixture (OMNi-BiOTiC STRESS) containing 9 human bacterial strains [Lactobacillus casei W56, Lactobacillus acidophilus W22, Lactobacillus paracasei W20, Bifidobacterium lactis W51 Bifidobacterium lactis W52, Lactobacillus salivarius W24, Lactococcus lactis W19, Lactobacillus plantarum W62, Bifidobacterium bifidum W23, with at least 7,5 billion CFU per one dose (3 g) and 15 billion CFU per two doses (6 g)] and vitamin B (B2, B6, B12), self-administered orally twice a day for 8 weeks
  Interventions: Dietary Supplement: Probiotic mixture (OMNi-BiOTiC STRESS)
- Placebo (Placebo Comparator): one powder portion bag self-administered orally twice a day for 8 weeks, identical in all aspects (organoleptic) as investigational product (IP) but containing excipient only.
  * Powder portion bags are suitable for participants with intolerance to yeasts or lactose
  * Each patient will receive a container with 112 powder portion bags (IP or placebo depending on the randomization) at the randomization period (0 weeks).
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic mixture (OMNi-BiOTiC STRESS) — OMNi-BiOTiC STRESS containing 9 human bacterial strains [Lactobacillus casei W56, Lactobacillus acidophilus W22, Lactobacillus paracasei W20, Bifidobacterium lactis W51, Bifidobacterium lactis W52, Lactobacillus salivarius W24, Lactococcus lactis W19, Lactobacillus plantarum W62, Bifidobacterium bifidum W23, with at least 7,5 billion CFU per one dose (3 g) and 15 billion CFU per two doses (6 g)] and vitamin B (B2, B6, B12),
  Arms: Probiotic
Other: Placebo — one powder portion bag self-administered orally twice a day for 8 weeks, identical in all aspects (organoleptic) as investigational product (IP) but containing excipient only.
  * Powder portion bags are suitable for participants with intolerance to yeasts or lactose
  * Each patient will receive a container with 112 powder portion bags (IP or placebo depending on the randomization) at the randomization period (0 weeks).
  Arms: Placebo

SUMMARY:
The objective of the current study is to evaluate the effect of a probiotic mixture on the adequate relief and faecal microbiota in obese patients with irritable bowel syndrome

DETAILED DESCRIPTION:
* The treatment period will last 8 weeks and after the treatment period, patients will be followed-up for another 2 weeks. Thus the overall trial period is the 10-week study period and end of 10th week is the end of the trial.
* Planned visits to gastroenterologists are at the screening period (-1 week), randomization period (0 weeks), and at the end of the treatment period (8th week).
* Patients will be instructed that unplanned visits to gastroenterologist are allowed only in case of a need or an urgency [e.g., adverse reactions, clinical deterioration and/or need for additional irritable bowel syndrome (IBS) management]. Unplanned visits will be recorded and does not exclude patients from the trial.
* For assessing other needed parameters (e.g., adequate relief, adverse reactions, irritable bowel syndrome (IBS) management) patients will be assessed by a physician, using an interactive voice response by telephone.
* Laboratory tests will be performed by certified clinical laboratories. Blood samples will be obtained by experienced trial nurses at the time of randomization (0 weeks).
* Anthropometric measurements will be assessed at the baseline and at the end of the treatment period (8th week).
* Irritable bowel syndrome (IBS) management (non-medication and medication therapy) will be assessed at the baseline, during the trial at the planned and unplanned visits to gastroenterologists, and at the end of the trial (by a physician using an interactive voice response by telephone). In a case of clinical deterioration IBS management is allowed during the trial and each will be recorded by gastroenterologists.
* Participants will receive 112 powder portion bags at the beginning of the trial and will be instructed to return the container after the 8-week treatment period. Leftover powder portion bags will be counted at the end of the treatment period (8th week) to estimate compliance. Compliant is considered a participant where no leftover powder portion bags will be recorded. Otherwise, the participant is considered non-compliant.
* Safety will be ensured by following adverse reactions during the trial. Scheduled assessment of adverse reactions is at the time of randomization, after 4 weeks, 8 weeks, and at the end of the trial. Responses will be recorded by a physician, at the planned visit of gastroenterologists and/or using an interactive voice response by telephone. Unscheduled recording of adverse reactions is during the entire trial by patients which will be instructed at the randomization period to report any adverse reactions to gastroenterologists using an interactive voice response by telephone. In a case of severe adverse reactions patients will be withdrawn from the trial and if needed. In case of a need or urgency (e.g., adverse reactions, clinical deterioration) clinical management will be provided in line with the best medical practice, by gastroenterologists and/or medical specialists depending on a medical condition.
* Patients can withdrawal from the trial any time. During the trial period withdrawal and its reason will be assessed by gastroenterologists at the visits or using an interactive voice response by telephone. Patients will be instructed in a case of a withdrawal to inform gastroenterologists and report the reason. In a lack of response the reason will be considered as other.

ELIGIBILITY:
Inclusion Criteria:

* Obese [Body mass index (BMI) ≥30] men or women with confirmed IBS (all subtypes based on Rome IV Diagnostic Criteria for IBS) aged between 18 and 65 years.
* Written informed consent.

Exclusion Criteria:

* Pregnancy or lactation
* Severe systemic illness [cancer, gastrointestinal illness (e.g., colitis, Crohn's disease, celiac disease, recurrent diverticulitis), chronic renal failure, an endocrine disorder, metabolic disorder, angina, congestive heart failure, uncontrolled hypertension] or severely impaired general health
* Organic abnormality which is excluded by full blood count, C-reactive protein or erythrocyte sedimentation rate, and thyroid-stimulating hormone for constipated IBS participants. To exclude other organic lower gastrointestinal disease faecal calprotectin will be checked, and celiac test and colonoscopy will be performed if needed.
* Previous abdominal surgery except for appendectomy, cholecystectomy and abdominal wall hernia repair
* History of psychiatric disorder
* History of participation in another clinical trial within 3 months before the onset of this trial
* Medications that could affect the outcomes: oral steroid, sulfasalazine, cholestyramine, misoprostol and probiotics usage 3 months prior to and during the study; and antacids with magnesium or aluminium usage during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Adequate relief | eight weeks
  Adequate relief (AR) related question of overall IBS symptoms "In the past 7 days have you had adequate relief of your IBS pain and discomfort?" which will be assessed weekly for 10 weeks (starting with 0 week till 10th week). A responder is defined as a patient who experiences AR (answers YES to AR related question) for at least 50% of the 10-week study period (5 of the 10 weekly assessments). 10-point analog scale will be used for the measurement of response rate among patients in each group.

SECONDARY OUTCOMES:
The fecal flora compositions | eight weeks
  The fecal flora compositions will be analyzed by Real Time polymerase chain reaction (PCR) for specific strain detection. The concordance rate of each patient's denaturing gradient gel electrophoresis (DGGE) profile before and after the treatment will be measured by the visual scale where each band of the DGGE profile represents a different organism and the similarity of band locations represents the same composition of the population of organisms.

OTHER OUTCOMES:
IBS Severity | eight weeks
  IBS severity will be assessed by the IBS symptom severity score (IBS SSS) questionnaire administered at the trial site by gastroenterologists and filled by patients at the time of randomization (0 weeks) and at the end of treatment (8th week). IBS-SSS consists of five items [abdominal pain, number of days with abdominal pain, bloating/distension, satisfaction with bowel habits, and IBS-related quality of life (QOL)], and each measure is rated from 0 to 100, with total scores ranging from 0 to 500. Participants with scores of <175, 175-300, and >300 are classified as mild, moderate, and severe groups.
IBS QOL | eight weeks
  IBS health related quality of life (QoL) will be assessed by IBS-36 questionnaire administered at the trial site by gastroenterologists and filled by patients at the time of randomization (0 week) and at the end of treatment (8th week). The IBS-36 consists of 36 questions scored on a 7-point Likert scale ranging from 0 through to 6, giving a maximal total score of 216. A final score is a sum of the scores of the 36 questions, with question 18 being reverse scored (i.e., for a patient score of 0, a score of 6 is entered). This instrument is negatively scored (i.e., a lower score equates to a better QoL) and assesses patients' symptoms over a last 2 months.
Psychological distress | eight weeks
  Psychological distress will be assessed by Hospital Anxiety and Depression Scale (HADS) questionnaire administered at the trial site by gastroenterologists and filled by patients at the time of randomization (0 week) and at the end of treatment (8th week). HADS is a 14-item scale with seven items each for anxiety and depression subscales. Scoring for each item ranges from zero to three. A subscale score >8 denotes anxiety or depression.

CONTACTS AND LOCATIONS:
Overall Officials: GORAN HAUSER, MD, PhD, Principal Investigator — KBC Rijeka; Medicinski fakultet Sveučilišta u Rijeci
Locations (2):
- Croatia (2):
  - Clinical Hospital Centre, Rijeka, Croatia
  - University Hospital Rijeka, Rijeka, Rijeka

IPD SHARING:
Plan to Share IPD: Yes
We will share all necessary documents which are not under GDPR protection
Supporting Information: Study Protocol, SAP, ICF
Time Frame: after enrollment, 50% of patients and will be available 6 months after study termination
Access Criteria: Patients, Ethic committee members, regulatory organisations
URL: https://hunm.eu/